CLINICAL TRIAL: NCT06472076
Title: A Randomized, Multicenter, Double-blind, Phase 3 Study to Investigate the Safety and Efficacy of Belrestotug in Combination With Dostarlimab Compared With Placebo in Combination With Pembrolizumab in Participants With Previously Untreated, Unresectable, Locally Advanced or Metastatic PD-L1 Selected Non-small Cell Lung Cancer (GALAXIES Lung-301)
Brief Title: A Study of Belrestotug Plus Dostarlimab Compared With Placebo Plus Pembrolizumab in Previously Untreated Participants With Programmed Death Ligand 1 (PD-L1) High Non-small-cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 213823
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Belrestotug; GSK4428859A; EOS-448; Dostarlimab; Pembrolizumab; PD-L1 selected NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dostarlimab; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dostarlimab plus belrestotug (Experimental)
  Interventions: Biological: Dostarlimab; Biological: Belrestotug
- Pembrolizumab plus placebo (Active Comparator)
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
  Arms: Dostarlimab plus belrestotug
Biological: Belrestotug — Belrestotug will be administered.
  Arms: Dostarlimab plus belrestotug
Biological: Pembrolizumab — Pembrolizumab will be administered.
  Arms: Pembrolizumab plus placebo
Drug: Placebo — Placebo will be administered.
  Arms: Pembrolizumab plus placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability profile of dostarlimab in combination with belrestotug when compared with pembrolizumab and placebo in participants with previously untreated, unresectable, locally advanced or metastatic PD-L1 high NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of locally advanced, unresectable NSCLC (not eligible for curative surgery and/or definitive radiotherapy with or without chemotherapy), or Metastatic NSCLC
* Has not received prior systemic therapy for their locally advanced or metastatic NSCLC.
* Provides a fresh tumor tissue sample obtained at the time of or after the initial diagnosis of locally advanced or metastatic NSCLC.
* Has a PD-L1-high (Tumor cells [TC] ≥50%) tumor
* Has measurable disease (at least 1 target lesion) based on RECIST 1.1
* Has an Eastern Cooperative Oncology Group (ECOG) Performance status (PS) score of 0 or 1.
* Has adequate organ function

Exclusion Criteria:

* Has NSCLC with a tumor that harbors any of the following molecular alterations:

  1. Epidermal growth factor receptor (EGFR) mutations that are sensitive to available targeted inhibitor therapy
  2. Anaplastic lymphoma kinase (ALK) translocations that are sensitive to available targeted inhibitor therapy
  3. Any other known genomic aberrations or oncogenic driver mutations for which a locally approved targeted therapy is available for first line treatment of locally advanced or metastatic NSCLC.
* Has had surgery within 4 weeks of the first dose of study intervention and has not recovered from AEs (i.e., has any ongoing surgery-related events ≥ Grade 1)/complications related to surgery or has received lung radiation therapy of >30 gray (Gy) within 6 months
* Has received prior therapy with any immune checkpoint inhibitors, including antibodies or drugs targeting PD-(L)1, Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), T cell immunoglobulin and ITIM domain (TIGIT), or other checkpoint pathways.
* Has never smoked, defined as smoking <100 tobacco cigarettes in a lifetime.
* Has an invasive malignancy or history of invasive malignancy other than the disease under study within the last 5 years, with the exception of those with a negligible risk of metastasis or death and/or treated with expected curative outcome.
* Has symptomatic, untreated, or actively progressin g brain metastases or leptomeningeal disease
* Has autoimmune disease or syndrome (current or history thereof) that required systemic treatment within the past 2 years.
* Has received any live vaccine within 30 days prior to first dose of study intervention.
* Has any history of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis.
* Has symptomatic ascites, pleural effusion, or pericardial effusion.
* Has active inflammatory bowel disease
* Has a history of significant acute or chronic cardiac diagnosis requiring intervention/treatment in the last 6 months.
* Has severe infection or complication thereof 4 weeks prior to randomisation including active tuberculosis.
* Has a history of allogeneic tissue/stem cell transplant or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to approximately 138 weeks
Number of Participants with TEAEs or SAEs leading to dose withdrawals or treatment discontinuation | Up to approximately 138 weeks

CONTACTS AND LOCATIONS:
Locations (112):
- United States (8):
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Olympia, Washington
- Argentina (9):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Florida
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
- Belgium (2):
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Mont Gaston
- Brazil (11):
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Belém
  - GSK Investigational Site, CuritibaPR
  - GSK Investigational Site, Florianópolis
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Londrina
  - GSK Investigational Site, Porto VelhoRondOnia
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, SAo JosE Do Rio PretoSP
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Bulgaria (2):
  - GSK Investigational Site, Haskovo
  - GSK Investigational Site, Plovdiv
- GSK Investigational Site, Halifax, Nova Scotia, Canada
- China (5):
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
- Finland (2):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Turku
- France (6):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
- GSK Investigational Site, Hamburg, Germany
- GSK Investigational Site, Shatin, Hong Kong
- India (10):
  - GSK Investigational Site, Gokul Shirgoan, Kolhapur
  - GSK Investigational Site, Ahmedabad-380016
  - GSK Investigational Site, Apex Wellness Hospital
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Bhubaneshwar
  - GSK Investigational Site, Bhubaneswar
  - GSK Investigational Site, Gūrgaon
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, New Delhi
- Japan (21):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Wakayama
- Mexico (4):
  - GSK Investigational Site, Guadajalara
  - GSK Investigational Site, La Paz BCS
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, San Luis Potosí City
- Netherlands (2):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Enschede
- Panama (2):
  - GSK Investigational Site, Panama City
  - GSK Investigational Site, Punta Pacifica Panama City Panama
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (16):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, BaracaldoVizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena Murcia
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valladolid
- GSK Investigational Site, Gävle, Sweden
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/